CLINICAL TRIAL: NCT03102060
Title: Gluten Free Diet for GVHD Prophylaxis
Brief Title: Gluten Free Diet in Preventing Graft Versus Host Disease in Patients Undergoing Donor Stem Cell Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roger Strair, MD, PhD, Associate Professor, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro20170000304; NCI-2017-00438 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 021701 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Graft Versus Host Disease; Hematopoietic Cell Transplantation Recipient
MeSH Terms: conditions — Graft vs Host Disease | interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (gluten free diet) (Experimental): Patients undergo a gluten free diet for 30 days during initial hospitalization for allo-SCT, from the time of admission to discharge.
  Interventions: Other: Dietary Intervention; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Dietary Intervention — Undergo gluten free diet
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies how well a gluten free diet works in preventing graft versus host disease in patients who are undergoing a donor stem cell transplant. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft versus host disease). A gluten free diet may decrease intestinal inflammation and graft versus host disease in patients who are undergoing a donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate and severity of gastrointestinal (GI) graft versus host disease (GVHD) in patients assigned to, and compliant with, a gluten free diet (GFD) during initial transplant hospitalization.

SECONDARY OBJECTIVES:

I. To determine the tolerance of, and compliance with, a GFD in patients undergoing allogeneic hematopoietic stem cell transplant (allo-SCT).

OUTLINE:

Patients undergo a gluten free diet for 30 days during initial hospitalization for allo-SCT, from the time of admission to discharge.

After completion of study, patients are followed up at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing an allo-SCT
* No history of celiac disease or non-celiac gluten sensitivity
* Male and female and all ethnic groups are eligible

Exclusion Criteria:

* Pregnant women
* Children are not eligible as the transplant program is certified as an adult only transplant program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Rate and severity of stage 2-4 GI acute (a)GVHD as determined by microbiome analysis of stool samples | Up to 12 months post allo-SCT
  To determine how often patients develop gastrointestinal graft-versus-host disease at various times after transplant
Rate and severity of all grade aGVHD and chronic GVHD as determined by microbiome analysis of stool samples | Up to 12 months post allo-SCT
  To determine what the severity is if graft-versus host disease develops.
Rate of compliance with GFD | Up to 30 days
  Adherence to diet will be recorded in a food diary. Compliance will be defined as > 67% of meals being gluten free.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States